CLINICAL TRIAL: NCT03226392
Title: A 12-week, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of QAW039 When Added to Standard-of-care Asthma Therapy in Patients With Uncontrolled Asthma
Brief Title: Study of Efficacy and Safety of QAW039 When Added to Standard-of-care Asthma Therapy in Patients With Uncontrolled Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQAW039A2317; 2017-001272-40 (EudraCT Number)
Record Dates: First submitted 2017-07-11; First posted 2017-07-21 (Actual); Results first posted 2020-02-28 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Asthma
Keywords: QAW039, uncontrolled asthma
MeSH Terms: conditions — Asthma | interventions — fevipiprant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- QAW039 (Active Comparator): QAW039 once daily
  Interventions: Drug: QAW039
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QAW039 — QAW039 once daily
  Arms: QAW039
Drug: Placebo — Placebo once daily
  Arms: Placebo

SUMMARY:
A randomized, multicenter, double-blind, placebo- controlled parallel-group study to determine the efficacy and safety of QAW039, compared with placebo, when added to standard-of-care (SoC) asthma therapy in adult and adolescent (≥ 12 years) patients with uncontrolled asthma with respect to change from baseline in forced expiratory volume in 1 second (FEV1) at the end of 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of asthma (according to GINA 2016) for a period of at least 6 months.
* Treated with medium dose inhaled corticosteroid (ICS), or high dose ICS, or low dose ICS plus long- acting beta agonist (LABA), or low dose ICS plus leukotriene receptor antagonist (LTRA), or medium dose ICS plus LABA for at least 3 months prior to Visit 1 and the doses have been stable for at least 4 weeks prior to Visit 1.
* FEV1 of ≤85% for patients aged ≥18 years. FEV1 of ≤90% for patients aged 12 to <18 years.
* Daytime asthma symptom score (0 to 6 scale) of ≥1 per day during 4 of the last 7 days of the placebo run- in period.
* Total daily SABA use ≥1 puff per day during 4 of the last 7 days of the placebo run-in period.
* Demonstrated reversible airway obstruction.
* Asthma control questionnaire (ACQ) score ≥ 1.5.

Exclusion Criteria:

* Use of other investigational drugs within 5 half-lives of enrollment, or within 30 days, whichever is longer.
* A resting QTcF (Fridericia) ≥450 msec (male) or

  ≥460 msec (female).
* Pregnant or nursing (lactating) women.
* Serious co-morbidities.
* Patients on >20 mg of simvastatin, > 40 mg of atorvastatin, >40 mg of pravastatin, or >2 mg of pitavastatin.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 704 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (134):
- United States (43):
  - Novartis Investigative Site, Andalusia, Alabama
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Newport Beach, California
  - Novartis Investigative Site, Rolling Hills Estates, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, San Jose, California
  - Novartis Investigative Site, Stockton, California
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Lafayette, Colorado
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Miami Gardens, Florida
  - Novartis Investigative Site, Tallahassee, Florida
  - Novartis Investigative Site, Winter Park, Florida
  - Novartis Investigative Site, Paducah, Kentucky
  - Novartis Investigative Site, Columbia, Maryland
  - Novartis Investigative Site, White Marsh, Maryland
  - Novartis Investigative Site, North Dartmouth, Massachusetts
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Rochester, Minnesota
  - Novartis Investigative Site, Saint Charles, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Warrensburg, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Brooklyn, New York
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Marion, Ohio
  - Novartis Investigative Site, Mayfield Heights, Ohio
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Altoona, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Mt. Pleasant, South Carolina
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, New Braunfels, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Murray, Utah
  - Novartis Investigative Site, Newport News, Virginia
  - Novartis Investigative Site, Spokane, Washington
- Brazil (7):
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, Porto Alegre, Porto Alegre RS
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Blumenau, Santa Catarina
  - Novartis Investigative Site, São Bernardo do Campo, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Sorocaba, São Paulo
- Bulgaria (4):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Rousse
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Stara Zagora
- Canada (3):
  - Novartis Investigative Site, Kingston, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Windsor, Ontario
- Colombia (4):
  - Novartis Investigative Site, Ibagué, Tolima Department
  - Novartis Investigative Site, Bogota DC
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Bucaramanga
- Germany (8):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lübeck
- Hungary (7):
  - Novartis Investigative Site, Hajdúnánás, HUN
  - Novartis Investigative Site, Kapuvár, HUN
  - Novartis Investigative Site, Püspökladány, HUN
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Siófok
  - Novartis Investigative Site, Szigetszentmiklós
- India (6):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Vadodara, Gujarat
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Bikaner, Rajasthan
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Dehradun, Uttarakhand
- Israel (4):
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Rehovot
- Italy (5):
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Milan
- Peru (6):
  - Novartis Investigative Site, Lima Cercado, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, San Martín de Porres, Lima region
  - Novartis Investigative Site, Cusco
  - Novartis Investigative Site, Lima
  - Novartis Investigative Site, Piura
- Novartis Investigative Site, San Juan, Puerto Rico
- Russia (11):
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, N.Novgorod
  - Novartis Investigative Site, Penza
  - Novartis Investigative Site, Perm
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Stavropol
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- South Korea (9):
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Bucheon-si, Gyeonggi-do
  - Novartis Investigative Site, Hwaseong-si, Gyeonggi-do
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Seoul
- Spain (9):
  - Novartis Investigative Site, Marbella, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Laredo, Cantabria
  - Novartis Investigative Site, Pozuelo de Alarcón, Madrid
  - Novartis Investigative Site, Barcelona, Vic
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Girona
  - Novartis Investigative Site, Santiago de Compostela
  - Novartis Investigative Site, Zaragoza
- Sweden (3):
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Umeå
  - Novartis Investigative Site, Visby
- Novartis Investigative Site, Bab Saadoun, Tunisia
- Vietnam (3):
  - Novartis Investigative Site, Haiphong
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=594
- See also: A Pediatric Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/ppatientsummary/ppatientsummaries?periodicPatientSummaryId=483

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from centers in Brazil (8), Bulgaria (4), Canada (3), Colombia (4), Germany (5), Hungary (7), India (5), Israel (5), Italy (4), Peru (6), Republic of Korea (5), Russian Federation (14), Spain (8), United States (36), Vietnam (3).
Groups:
- QAW039: QAW039 150mg once daily
Period: Overall Study
Arm/Group | QAW039 | Placebo
Started | 352 | 352
FAS | 352 | 350 (2 patients in the placebo were mis-randomized, not treated, not included due to "technical problems)
Completed | 341 | 344
Not Completed | 11 | 8
Not completed — Protocol Deviation | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Technical Problems | 0 | 2
Not completed — Subject/Guardian Decision | 7 | 6

BASELINE CHARACTERISTICS:
Population: Two patients were randomized in error (mis-randomized) and did not receive any study drug; for these patients the reason for discontinuation is given as "technical problems"
Groups:
- Total: Total of all reporting groups
Arm/Group | QAW039 | Placebo | Total
Number analyzed (Participants) | 352 | 350 | 702
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Two patients in the placebo group were randomized in error and did not receive any study drug; for these patients the reason for discontinuation is given as "technical problems"
  Years | 50.4 (14.87) | 50.2 (14.39) | 50.3 (14.62)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two patients in the placebo group were randomized in error and did not receive any study drug; for these patients the reason for discontinuation is given as "technical problems"
  Participants
    Female | 216 | 218 | 434
    Male | 136 | 132 | 268
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Two patients in the placebo group were randomized in error and did not receive any study drug; for these patients the reason for discontinuation is given as "technical problems"
  Participants
    Black | 26 | 18 | 44
    Asian | 41 | 46 | 87
    Native American | 12 | 12 | 24
    Pacific Islander | 2 | 0 | 2
    Other | 55 | 58 | 113
    Caucasian | 216 | 216 | 432

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pre-dose FEV1
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Baseline is defined as the last available FEV1 measurement taken prior to the first dose of randomized study drug.
Time Frame: Baseline and Week 12
Population: Full Analysis Set (FAS): all randomized patients who received at least one dose of study medication. Patients in the FAS were analyzed according to the treatment they were assigned to at randomization.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QAW039 | Placebo
Number analyzed (Participants) | 352 | 350
Liters | 0.126 (0.00177) | 0.157 (0.0177)
Statistical Analysis 1: Comparison: QAW039 vs Placebo; Test type: Superiority; p = 0.214, ANCOVA; Mean Difference (Net) = -0.031, 95% CI 2-sided [-0.080 to 0.018]

2. Secondary Outcome: Change From Baseline in Daytime Asthma Symptom Score
Description: Daytime asthma symptoms are evaluated through four questions and each of them will be rated on a scale of 0 to 6. Higher scores indicate more severe asthma-related symptoms. A mean score is calculated for the responses to 4 questions.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | QAW039 | Placebo
Number analyzed (Participants) | 352 | 350
Score | -0.55 (0.034) | -0.45 (0.034)
Statistical Analysis 1: Comparison: QAW039 vs Placebo; Test type: Superiority; p = 0.035, ANCOVA; Mean Difference (Net) = -0.10, 0.035% CI 2-sided [-0.19 to 0.01]

3. Secondary Outcome: Change From Baseline in Number of Puffs of SABA Taken Per Day
Description: Daily use of SABA (the number of rescue medication puffs taken in the previous 12 hours) was recorded using a patient electronic diary (referred to as eDiary or eDiary/ePEF). Patients were instructed to routinely complete the patient diary twice daily - at the same time each morning and each evening, approximately 12 hours apart.
Time Frame: Baseline (daily mean for up to three weeks prior to baseline visit) and Week 12 (daily mean post baseline up to Week 12)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs per day
Arm/Group | QAW039 | Placebo
Number analyzed (Participants) | 352 | 350
Puffs per day | -0.89 (0.066) | -0.88 (0.066)
Statistical Analysis 1: Comparison: QAW039 vs Placebo; Test type: Superiority; p = 0.893, ANCOVA; Mean Difference (Net) = 0.093, 95% CI 2-sided [-0.20 to 0.17]

4. Secondary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire for 12 Years and Older (AQLQ+12) Score
Description: AQLQ is a 32-item instrument administered as a self-assessment. AQLQ+12 is a modified version of AQLQ developed to measure functional impairments of participants aged 12-70 years. It is divided into 4 domains: activity limitation, symptoms, emotional function, and environmental stimuli. Participants were asked to recall their experiences during the last 2 weeks and respond to each question on a 7-point scale (1=severe impairment, 7=no impairment), where higher scores indicated "better quality of life." Overall AQLQ+12 score is the mean of all 32 responses.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | QAW039 | Placebo
Number analyzed (Participants) | 352 | 350
units on a scale | 0.77 (0.043) | 0.72 (0.043)
Statistical Analysis 1: Comparison: QAW039 vs Placebo; Test type: Superiority; p = 0.448, ANCOVA; Mean Difference (Net) = 0.061, 95% CI 2-sided [-0.07 to 0.17]

ADVERSE EVENTS:
Time Frame: After signing informed consent to 30 days after last dose, assessed up to 16 weeks.
Groups:
- QAW039 150 mg: QAW039 150 mg
- Placebo: Placebo
Arm/Group | QAW039 150 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/352 | 0/350
Serious Adverse Events (participants affected / at risk) | 7/352 | 3/350
Other Adverse Events (participants affected / at risk) | 94/352 | 116/350
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QAW039 150 mg (N=352) | Placebo (N=350)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QAW039 150 mg (N=352) | Placebo (N=350)
Bronchitis (Infections and infestations) | 9 | 6
Influenza (Infections and infestations) | 4 | 1
Nasopharyngitis (Infections and infestations) | 10 | 24
Pharyngitis (Infections and infestations) | 5 | 2
Respiratory tract infection viral (Infections and infestations) | 5 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 10
Upper respiratory tract infection bacterial (Infections and infestations) | 3 | 6
Viral upper respiratory tract infection (Infections and infestations) | 12 | 8
Contusion (Injury, poisoning and procedural complications) | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 7
Headache (Nervous system disorders) | 5 | 14
Asthma (Respiratory, thoracic and mediastinal disorders) | 46 | 61
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT03226392/Prot_001.pdf
  • Statistical Analysis Plan (2019-08-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT03226392/SAP_000.pdf